CLINICAL TRIAL: NCT03976960
Title: Prospective, Multicenter, Clinical and Biological Database Set-up in Colon Cancer and Colic Tumors
Brief Title: Clinical and Biological Database in Colon Cancer and Colic Tumors
Acronym: BCBCOLON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BCB2014/01
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Cancer Colon
Keywords: cancer; colon; tumor; colic
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms; Colic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological collection (Experimental): For all the patients include in the study :
  samples of blood samples collected before or after surgery but also samples in paraffin-embedded tissue sections.
  In parallel to this biological collection, standardized clinical data will be entered into a database
  Interventions: Other: Biological collection

INTERVENTIONS:
Other: Biological collection — The biological collection will also include samples of blood samples collected before or after surgery but also samples frozen and/or paraffin-embedded tissue sections.

SUMMARY:
Developement of a clinical and biological database in colon cancer and colic tumors in order to better understand tumor invasion and metastatic scattering processes. The investigators hope that a better understanding of tumoral invasion process will lead to the discovery of new biomarkers and new drugs.

DETAILED DESCRIPTION:
As the second leading cause of cancer-related death in France, colorectal cancer is a major public health problem. Each year, 37 000 cases are newly diagnosed in France and 17 000 patients die of the disease.

Colorectal cancer is due to molecular and genetic damages involved in all tumorigenesis steps, transition from healthy tissue to adenoma and finally to invasive carcinoma stage. The investigators hope that a to better understand tumor invasion and metastatic scattering processes will allow therapeutic innovation and the emergence of new biomarkers.

However, the study of early tumorigenesis phases as well as advanced stages of the disease is currently limited due to a lack of tissue samples.

In this context, the Montpellier Cancer Institute (ICM) decided to initiate a biological collection dedicated to the tissular and blood samples of patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient undergoing colon cancer surgery (stage I, II, III and IV)
2. Patient operated for liver or lung or peritoneal carcinomatosis metastases originating from colon cancer
3. Patient operated for pre-neoplastic lesion (adenomatous polyp /villous adenoma polyp),
4. Patient with familial polyposis eligible for colectomy
5. Age > 18 years
6. Signed informed consent

Exclusion Criteria:

1. Patient not affiliated to Social Protection system
2. Patient unable to understand or comply with study instructions or requirements for psychological, family, social or geographical reasons
3. Patient under guardianship
4. Minor patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of clinical risk factors for colorectal cancer | Until the study completion : 6 years
Number of biological risk factors for colorectal cancer | Until the study completion : 6 years

CONTACTS AND LOCATIONS:
Overall Officials: ERIC ASSENAT, M.D, Study Chair — Institut régional du cancer de Montpellier
Locations (2):
- France (2):
  - CHRU de Montpellier, Montpellier, Hérault
  - Institut Régional du cancer de Montpellier, Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National estimate of cancer incidence and mortality in France between 1980 and 2012. — https://www.google.com/search?client=firefox-b-d&sxsrf=ALeKk0251JuQRT2bZiWL8ut7KwGhX0TKeQ:1596454499279&q=Estimation+nationale+de+l%27incidence+et+de+la+mortalit%C3%A9+par+cancer+en+France+entre+1980+et+2012.+Partie+1-+Tumeurs+solides.+Traitement+:+INCA+2013.&spell=1&sa=X&ved=2ahUKEwj7lNG6-P7qAhVKxIUKHZeSCMMQBSgAegQICxAq&biw=1920&bih=1006